CLINICAL TRIAL: NCT05119829
Title: Melanoma: Genomic Profiles, Molecular Markers and Therapeutic Implications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: Gen_Melanoma_HeCOG
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-Fixed-Paraffin-Embedded (FFPE) tumor tissue blocks will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate the genomic profiles and investigate the prevalence of germ line and pathogenic mutations in Greek population with early and metastatic melanoma and their correlation with the treatment and prognosis of the disease.

DETAILED DESCRIPTION:
In this context, it is aimed to utilize tissue biopsy tests that will focus on specific areas of clinical applications, namely, diagnosis, prognosis and identification of mutations for targeted therapy and assessment of acquiring treatment resistance. Thus, the tissue biopsy Next Generation Sequencing (NGS) panels in development by NIPD Genetics will be used in clinical practice as complementary diagnostics.

For tumor genotyping of the 200 patients with melanoma skin cancer in the present study it will be used the comprehensive tissue biopsy melanoma cancer panel from NIPD Genetics These panels are designed to target clinically actionable and clinically significant mutations that will provide physicians with genetic information regarding a) prediction of the patient's response to targeted therapy, b) prognosis, that is, prediction of clinical outcome, c) diagnosis and molecular classification of melanoma cancer. The panel allows for the detection of single nucleotide (SNVs) and copy number variants (CNVs), as well as gene fusions and indels; it necessitates at least 400ng of appropriate quality DNA template that is achievable from FFPE samples and is validated with molecular standards and controls for the exclusion of artefacts.

Thorough histological evaluation of the Formalin-Fixed-Paraffin-Embedded (FFPE) tumor tissue blocks will be done by an experienced pathologist to evaluate H&E sections for confirmation of diagnosis, histologic type, grade and tumor cell content (TCC%). DNA isolation will be performed from 10 μm whole sections following manual macro-dissection to enrich samples for tumor DNA, whereby TCC will be assessed as an approximate metric for tumor DNA in the extracted samples, corresponding to tumor nuclei vs. all nuclei in the areas marked for macro-dissection.

A total of 200 patients with melanoma skin cancer are expected to be included in the analysis based on the number of patients registered in the Hellenic Cooperative Oncology Group's (HeCOG's) database along with the ability to achieve precision around the primary and secondary endpoints. Primary endpoint will be the evaluation of the prevalence of mutations, while the secondary endpoint will be the assessment of prognostic significance of mutations with respect to overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Melanoma skin cancer patients
* the ability to achieve FFPE

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed melanoma skin cancer. Patients are treated in Hellenic Cooperative oncology Group affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 1998-02-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of prevalence mutation | January 2022 to September 2022
  Evaluation of prevalence mutation

SECONDARY OUTCOMES:
ognostic significance of mutations with respect to overall survival | January 2022 to September 2022
  assessment of prognostic significance of mutations with respect to overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Dept of Medical Oncology, Metropolitan Hospital, Athens, Greece

REFERENCES:
- [Background] Forsea AM, Del Marmol V, Stratigos A, Geller AC. Melanoma prognosis in Europe: far from equal. Br J Dermatol. 2014 Jul;171(1):179-82. doi: 10.1111/bjd.12923. Epub 2014 Jun 24. PMID 24588115
- [Background] Khair DO, Bax HJ, Mele S, Crescioli S, Pellizzari G, Khiabany A, Nakamura M, Harris RJ, French E, Hoffmann RM, Williams IP, Cheung A, Thair B, Beales CT, Touizer E, Signell AW, Tasnova NL, Spicer JF, Josephs DH, Geh JL, MacKenzie Ross A, Healy C, Papa S, Lacy KE, Karagiannis SN. Combining Immune Checkpoint Inhibitors: Established and Emerging Targets and Strategies to Improve Outcomes in Melanoma. Front Immunol. 2019 Mar 19;10:453. doi: 10.3389/fimmu.2019.00453. eCollection 2019. PMID 30941125
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Hodi FS, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Cowey CL, Lao CD, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hill A, Hogg D, Marquez-Rodas I, Jiang J, Rizzo J, Larkin J, Wolchok JD. Nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone in advanced melanoma (CheckMate 067): 4-year outcomes of a multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1480-1492. doi: 10.1016/S1470-2045(18)30700-9. Epub 2018 Oct 22. PMID 30361170
- [Background] Hayward NK, Wilmott JS, Waddell N, Johansson PA, Field MA, Nones K, Patch AM, Kakavand H, Alexandrov LB, Burke H, Jakrot V, Kazakoff S, Holmes O, Leonard C, Sabarinathan R, Mularoni L, Wood S, Xu Q, Waddell N, Tembe V, Pupo GM, De Paoli-Iseppi R, Vilain RE, Shang P, Lau LMS, Dagg RA, Schramm SJ, Pritchard A, Dutton-Regester K, Newell F, Fitzgerald A, Shang CA, Grimmond SM, Pickett HA, Yang JY, Stretch JR, Behren A, Kefford RF, Hersey P, Long GV, Cebon J, Shackleton M, Spillane AJ, Saw RPM, Lopez-Bigas N, Pearson JV, Thompson JF, Scolyer RA, Mann GJ. Whole-genome landscapes of major melanoma subtypes. Nature. 2017 May 11;545(7653):175-180. doi: 10.1038/nature22071. Epub 2017 May 3. PMID 28467829
- [Background] Shain AH, Joseph NM, Yu R, Benhamida J, Liu S, Prow T, Ruben B, North J, Pincus L, Yeh I, Judson R, Bastian BC. Genomic and Transcriptomic Analysis Reveals Incremental Disruption of Key Signaling Pathways during Melanoma Evolution. Cancer Cell. 2018 Jul 9;34(1):45-55.e4. doi: 10.1016/j.ccell.2018.06.005. PMID 29990500
- [Background] Long GV, Menzies AM, Nagrial AM, Haydu LE, Hamilton AL, Mann GJ, Hughes TM, Thompson JF, Scolyer RA, Kefford RF. Prognostic and clinicopathologic associations of oncogenic BRAF in metastatic melanoma. J Clin Oncol. 2011 Apr 1;29(10):1239-46. doi: 10.1200/JCO.2010.32.4327. Epub 2011 Feb 22. PMID 21343559
- [Background] Carlino MS, Haydu LE, Kakavand H, Menzies AM, Hamilton AL, Yu B, Ng CC, Cooper WA, Thompson JF, Kefford RF, O'Toole SA, Scolyer RA, Long GV. Correlation of BRAF and NRAS mutation status with outcome, site of distant metastasis and response to chemotherapy in metastatic melanoma. Br J Cancer. 2014 Jul 15;111(2):292-9. doi: 10.1038/bjc.2014.287. Epub 2014 Jun 10. PMID 24918823
- [Background] Shain AH, Bastian BC. From melanocytes to melanomas. Nat Rev Cancer. 2016 Jun;16(6):345-58. doi: 10.1038/nrc.2016.37. Epub 2016 Apr 29. PMID 27125352
- [Background] Long GV, Weber JS, Infante JR, Kim KB, Daud A, Gonzalez R, Sosman JA, Hamid O, Schuchter L, Cebon J, Kefford RF, Lawrence D, Kudchadkar R, Burris HA 3rd, Falchook GS, Algazi A, Lewis K, Puzanov I, Ibrahim N, Sun P, Cunningham E, Kline AS, Del Buono H, McDowell DO, Patel K, Flaherty KT. Overall Survival and Durable Responses in Patients With BRAF V600-Mutant Metastatic Melanoma Receiving Dabrafenib Combined With Trametinib. J Clin Oncol. 2016 Mar 10;34(8):871-8. doi: 10.1200/JCO.2015.62.9345. Epub 2016 Jan 25. PMID 26811525
- [Background] Catalanotti F, Cheng DT, Shoushtari AN, Johnson DB, Panageas KS, Momtaz P, Higham C, Won HH, Harding JJ, Merghoub T, Rosen N, Sosman JA, Berger MF, Chapman PB, Solit DB. PTEN Loss-of-Function Alterations Are Associated With Intrinsic Resistance to BRAF Inhibitors in Metastatic Melanoma. JCO Precis Oncol. 2017 Jun 23;1:PO.16.00054. doi: 10.1200/PO.16.00054. eCollection 2017. PMID 32913971
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2016 Mar 24;165(1):35-44. doi: 10.1016/j.cell.2016.02.065. Epub 2016 Mar 17. PMID 26997480
- [Background] Whiteman DC, Baade PD, Olsen CM. More people die from thin melanomas (⩽1 mm) than from thick melanomas (>4 mm) in Queensland, Australia. J Invest Dermatol. 2015 Apr;135(4):1190-1193. doi: 10.1038/jid.2014.452. Epub 2014 Oct 20. No abstract available. PMID 25330295
- [Background] D'Angelo SP, Larkin J, Sosman JA, Lebbe C, Brady B, Neyns B, Schmidt H, Hassel JC, Hodi FS, Lorigan P, Savage KJ, Miller WH Jr, Mohr P, Marquez-Rodas I, Charles J, Kaatz M, Sznol M, Weber JS, Shoushtari AN, Ruisi M, Jiang J, Wolchok JD. Efficacy and Safety of Nivolumab Alone or in Combination With Ipilimumab in Patients With Mucosal Melanoma: A Pooled Analysis. J Clin Oncol. 2017 Jan 10;35(2):226-235. doi: 10.1200/JCO.2016.67.9258. Epub 2016 Nov 7. PMID 28056206
- [Background] Stratton MR, Campbell PJ, Futreal PA. The cancer genome. Nature. 2009 Apr 9;458(7239):719-24. doi: 10.1038/nature07943. PMID 19360079
- [Background] Chin L, Gray JW. Translating insights from the cancer genome into clinical practice. Nature. 2008 Apr 3;452(7187):553-63. doi: 10.1038/nature06914. PMID 18385729
- [Background] Forbes SA, Beare D, Boutselakis H, Bamford S, Bindal N, Tate J, Cole CG, Ward S, Dawson E, Ponting L, Stefancsik R, Harsha B, Kok CY, Jia M, Jubb H, Sondka Z, Thompson S, De T, Campbell PJ. COSMIC: somatic cancer genetics at high-resolution. Nucleic Acids Res. 2017 Jan 4;45(D1):D777-D783. doi: 10.1093/nar/gkw1121. Epub 2016 Nov 28. PMID 27899578
- [Background] Cancer Genome Atlas Research Network; Weinstein JN, Collisson EA, Mills GB, Shaw KR, Ozenberger BA, Ellrott K, Shmulevich I, Sander C, Stuart JM. The Cancer Genome Atlas Pan-Cancer analysis project. Nat Genet. 2013 Oct;45(10):1113-20. doi: 10.1038/ng.2764. PMID 24071849
- [Background] Landrum MJ, Lee JM, Riley GR, Jang W, Rubinstein WS, Church DM, Maglott DR. ClinVar: public archive of relationships among sequence variation and human phenotype. Nucleic Acids Res. 2014 Jan;42(Database issue):D980-5. doi: 10.1093/nar/gkt1113. Epub 2013 Nov 14. PMID 24234437
- [Background] NCCN Clinical Practice Guidelines in Oncology TM. 2009
- [Background] Jennings LJ, Arcila ME, Corless C, Kamel-Reid S, Lubin IM, Pfeifer J, Temple-Smolkin RL, Voelkerding KV, Nikiforova MN. Guidelines for Validation of Next-Generation Sequencing-Based Oncology Panels: A Joint Consensus Recommendation of the Association for Molecular Pathology and College of American Pathologists. J Mol Diagn. 2017 May;19(3):341-365. doi: 10.1016/j.jmoldx.2017.01.011. Epub 2017 Mar 21. PMID 28341590
- [Background] Koumbaris G, Kypri E, Tsangaras K, Achilleos A, Mina P, Neofytou M, Velissariou V, Christopoulou G, Kallikas I, Gonzalez-Linan A, Benusiene E, Latos-Bielenska A, Marek P, Santana A, Nagy N, Szell M, Laudanski P, Papageorgiou EA, Ioannides M, Patsalis PC. Cell-Free DNA Analysis of Targeted Genomic Regions in Maternal Plasma for Non-Invasive Prenatal Testing of Trisomy 21, Trisomy 18, Trisomy 13, and Fetal Sex. Clin Chem. 2016 Jun;62(6):848-55. doi: 10.1373/clinchem.2015.252502. Epub 2016 Apr 26. PMID 27117469